CLINICAL TRIAL: NCT03916679
Title: Safety and Effectiveness of MESO-CAR T Cells Therapy for Relapsed and Refractory Epithelial Ovarian Cancer
Brief Title: MESO-CAR T Cells Therapy for Relapsed and Refractory Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MESO-OS
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; CAR-T; MESO; Relapsed and Refractory
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-MESO CAR-T cells (Experimental): Administration with anti-MESO CAR-T cells in the MESO-positive ovarian cancer patients
  Interventions: Biological: anti-MESO CAR-T cells

INTERVENTIONS:
Biological: anti-MESO CAR-T cells — Retroviral vector-transduced autologous T cells to express anti-MESO CARs
  Other Names: Fludarabine 30mg/m2/d; Cyclophosphamide 300mg/m2/d

SUMMARY:
The goal of this clinical trial is to study the feasibility and efficacy of anti-MESO antigen receptors (CARs) T cell therapy for relapsed and refractory epithelial ovarian cancer.

DETAILED DESCRIPTION:
Primary Objectives

To determine the feasibility ad safety of anti-MESO CAR-T cells in treating patients with MESO-positive ovarian cancer.

Secondary Objectives

To access the efficacy of anti-MESO CAR-T cells in patients with ovarian cancer.

To determine in vivo dynamics and persistency of anti- MESO CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

- 18 to 70 Years Old, female; Expected survival > 12 weeks; Clinical performance status of ECOG score 0-2; Patients who have previously been treated with second- line or more lines of standard treatment are not effective (No remission or recurrence after remission); At least one measurable tumor foci according to RECIST standard 1.1 ; Positive Mesothelin expression in tumor tissues; Creatinine ≤ 1.5×ULN; ALT and AST ≤ 3×ULN; Total bilirubin ≤ 2×ULN; Hemoglobin≥90g/L; Absolute counting of neutrophils≥1000uL ; Absolute counting of lymphocytes>0.7×10^9/L; Counting of Platelet≥75000/uL; The venous access required for collection can be established without contraindications for leukocyte collection; Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

- Accompanied by other uncontrolled malignant tumors; Active hepatitis B, hepatitis C, syphilis, HIV infection; Suffering severe cardiovascular or respiratory disease; Any other diseases could affect the outcome of this trial; Any affairs could affect the safety of the subjects or outcome of this trial; Pregnant or lactating women, or patients who plan to be pregnancy during or after treatment; There are active or uncontrollable infections (except simple urinary tract infections or upper respiratory tract infections) that require systemic therapy 14 days or 14 days prior to assignment; Patients who are accounted by researchers to be not appropriate for this test; Received CAR-T treatment or other gene therapies before assignment; Subject suffering disease affects the understanding of informed consent or comply with study protocol.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-20 (Estimated); Primary Completion 2022-04-20 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 12 months post infusion

SECONDARY OUTCOMES:
Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm | 12 months post infusion
Progress Free Survival (PFS) after administration | 12 months post infusion
Duration of CAR-positive T cells in circulation | 12 months post infusion
Detection of PD1 antibody in serum | 12 months post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jianwei Zhou, M.D., Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided